CLINICAL TRIAL: NCT00183950
Title: Phase I/II Study of Noscapine for Patients With Low Grade Non Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia Refractory to Chemotherapy
Brief Title: Study of Noscapine for Patients With Low Grade Non Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia Refractory to Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-99-16
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Noscapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Noscapine

SUMMARY:
This study is for patients with non-hodgkin's lymphoma or chronic lymphocytic leukemia, which has failed to shrink or has returned after previous treatment with chemotherapy. The purpose of this study is to find out whether patients with these types of cancer will have their tumor shrunk after treatment with a drug called Noscapine. The second purpose is to see what are the side effects of this drug. This drug is being used as an over-the-counter cough suppressor in Europe and Japan, but has also shown to be effective against cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low grade NHL (follicular lymphoma, small cell lymphocytic lymphoma, marginal cell lymphoma, monocytoid B-cell lymphoma, MALT lymphoma, plasmacytoid lymphocytic lymphoma) or chronic lymphocytic leukemia who have demonstrated chemotherapy resistance (have not achieved CR,CRu, PR)or who have relapsed at any time following a response (CR, CRu, PR) after at least one therapy regimen, including chemotherapy, Rituximab, or high dose chemotherapy with stem cell rescue.
* Karnofsky performance status 60 % or greater.
* Creatinine less or equal to 2.0 mg/dl, bilirubin less or equal to 2.0 mg/dl, SGPT/SGOT less or equal to 4 x upper normal range

Exclusion Criteria:

* Patients with unconfirmed complete response(CRu)after last treatment and who currently remain in CRu.
* Pregnant or lactating women.
* Disease-specific treatment less than 1 month prior to starting this study.
* CNS disease.
* HIV-positive patients.
* Other cancer, except basal cell or squamous cell cancer of the skin or carcinoma in-situ of cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States